CLINICAL TRIAL: NCT05226364
Title: Effect of Tourniquet Abstention on Pain Reduction in Venous Sampling in the Elderly People : Randomized Trial
Brief Title: Effect of Tourniquet Abstention on Pain Reduction in Venous Sampling in the Elderly People
Acronym: NO-GARROT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHRD0319; 2021-A02936-35 (Other: ID-RCB)
Record Dates: First submitted 2021-12-15; First posted 2022-02-07 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Venous Puncture
Keywords: Venous Puncture; Tourniquet; Pain; Elderly people
MeSH Terms: conditions — Pain | interventions — Tourniquets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rubber tourniquet (Experimental): The blood sample is taken with a rubber tourniquet,
  Interventions: Procedure: Rubber tourniquet
- Fabric tourniquet (Experimental): The blood sample is taken with a a fabric tourniquet
  Interventions: Procedure: Fabric tourniquet
- No tourniquet (Experimental): The blood sample is taken without tourniquet
  Interventions: Procedure: Without tourniquet

INTERVENTIONS:
Procedure: Rubber tourniquet — The blood sample is taken with a rubber tourniquet
  Arms: Rubber tourniquet
Procedure: Fabric tourniquet — The blood sample is taken with a fabric tourniquet
  Arms: Fabric tourniquet
Procedure: Without tourniquet — The blood sample is taken without tourniquet
  Arms: No tourniquet

SUMMARY:
This prospective study evaluates the effect of abstaining from tourniquets on pain reduction during the venous puncture of the elderly people.

DETAILED DESCRIPTION:
Almost 3 million people aged 70 and over are hospitalized once or more each year. The implementation of multiple treatments in these fragile patients, often poly-pathological requires a regular biological monitoring. For these patients, samples must be taken on average every two days.

This population often has a fragile venous capital due to reduced skin elasticity, undernutrition more or less associated with dehydration, the use of certain venous-toxic treatments and / or repetition of the gesture taking into account the monitoring biological closely related to long-term therapies.

With the aim of well-treatment and well-being, the reduction of patient pain is one of the major concerns of caregivers and in particular pain induced by treatment.

In children, the practice of harvesting without tourniquet is already frequent (18) and our preliminary study has confirmed us on the tourniquet as one of the acts responsible for the pain that the caregiver can possibly abstain.

No study had been conducted on this subject in the adult population and more particularly the elderly population. This prospective study evaluates the effect of abstaining from tourniquets on pain reduction during the venous puncture of the elderly people.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 75 years and over,
* Hospitalized in internal medicine or geriatric department,
* For which the 2 upper limbs are accessible to venous puncture (due to the multiple attempts that may be necessary to take a sample during the hospitalization),
* For which at least one vein is visible or palpable on an upper limb,
* Without venous puncture since admission in the department,
* Patient who did not receive a topical anesthetic before the venous puncture (Emla type)
* Communicating patient, able to assess their pain on a digital scale,
* Patients with affiliation to a social security system or beneficiary ,
* Written informed consent (IC) obtained.

Exclusion Criteria:

* Patient already included,
* Previous pain localized to the upper limbs,
* Hematoma at the planned site of skin-vascular breakage,
* Hemiplegic or quadriplegic patient,
* Patient with lymphedema in the upper limbs,
* Patient with behavioral disorders that may interfere with the proper functioning of the sampling,
* Patient with cognitive impairment preventing understanding of the study and adequate assessment pain (CODEX cognitive score of category C or D),
* Patient placed under legal protection (guardianship).

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Comparison of the maximum pain associated with venous puncture, in elderly patients with a visible or palpable vein depending on the method of sampling. | At the end of the study, an average of 12 month
  Assessment of maximum pain on examination (including pain from skin-vascular invasion and tourniquet pain)by the patient using a verbal numerical scale (EN) rated from 0 to 10.
  This measure concerns the 1st sampling as a whole, regardless of the number of attempts necessary to obtain it and their terms

SECONDARY OUTCOMES:
Proportion of elderly patients with a visible or palpable vein | At the end of the study, an average of 12 month
  Estimate of the proportion of patients corresponding to phlebological prerequisites of the study (vein visible or palpable on at least one of the two upper limbs) on all elderly people meeting the other selection criteria upon admission to the service for the duration of the research
Comparison of the number of cutaneous-vascular breaks necessary for obtain a blood sample, according to the venous sampling procedure | At the end of the study, an average of 12 month
  Compilation of the number of cutaneous-vascular ruptures performed until obtention of a sample sent to laboratory
Comparison of the time taken to obtain a blood sample by caregivers, according to the venous sampling procedures | At the end of the study, an average of 12 month
  Measurement of the time required for this sample using timing from the moment the nurse is ready and until the end of the filling of the first tube sampled. This timing is performed by the caregiver himself and not by the third party who will collect the patient's pain and who is not present, in order to avoid any external influence linked to the performance of the gesture during the evaluation of the main criterion
Comparison of the ease of taking the sample by caregivers, according to the venous sampling procedure | At the end of the study, an average of 12 month
  Collection of the ease of performing the sampling by the caregivers via a Likert-type question (very easy, rather easy, rather difficult, very difficult) filled in after each sampling.
  In addition, the need to change arms or to call on another caregiver to perform the procedure will be noted.
Estimation of the pain due to the tourniquet and to the cutaneous-vascular breaks in patients where sample was taken with tourniquet | At the end of the study, an average of 12 month
  Verbal numerical scale measurements of tourniquet pain and pain due to vascular break (groups with tourniquet only).
  0 = No pain, 5 = moderate pain and 10 = Worst possible pain.
Comparison of the frequency of side effects: malaise, hematoma at the cutaneous-vascular break site, according to the venous sampling procedure ; hematoma and / or skin abrasion at the tourniquet, in patients collected with tourniquet | At the end of the study, an average of 12 month
  The presence of hematoma (s) will be observed in each group the next day of the sample by a caregiver separate from the one who performed the sample. The caregiver will also note the presence of skin abrasions related to possible use of tourniquet. Other unwanted events will also be collected, in particular: vagal unease during or after the sample, hemorrhage, ...
Comparison of the frequency of hemolysis of the sample, according to the venous sampling procedure | At the end of the study, an average of 12 month
  Proportion of samples having to be carried out again for hemolysis
Estimation of the influence of the nurse's experience on the efficiency of venous sampling on the duration of blood collection | At the end of the study, an average of 12 month
  Estimation of the effect of the mode of venipuncture (arm), according to the experience of the nurse on the duration of blood collection.
  The duration of the blood sampling is expressed in minute.
Estimation of the influence of the nurse's experience on the efficiency of venous sampling on pain | At the end of the study, an average of 12 month
  Estimation of the effect of the mode of venipuncture (arm), according to the experience of the nurse on pain.
  Verbal numerical scale measurements was used : 0 = No pain, 5 = moderate pain and 10 = Worst possible pain.
Estimation of the influence of the type of material used on the efficiency of venous sampling on pain | At the end of the study, an average of 12 month
  Estimation of the effect of the mode of venipuncture (arm), according to the type of material (butterfly needle, diameter) on pain.
  Verbal numerical scale measurements was used : 0 = No pain, 5 = moderate pain and 10 = Worst possible pain.
Estimation of the influence of the type of material used on the efficiency of venous sampling on the duration of blood collection | At the end of the study, an average of 12 month
  Estimation of the effect of the mode of venipuncture (arm), according to the type of material (butterfly needle, diameter) on the duration of blood collection.
  The duration of the blood sampling is expressed in minute.
Frequency of failures (regardless of the venous sampling method used) and refusal of the sample venous without tourniquet | At the end of the study, an average of 12 month
  Number of failures (regardless of the venous sampling method used) and refusal of the sample venous without tourniquet

CONTACTS AND LOCATIONS:
Overall Officials: Vella QUILLIEN, Principal Investigator — Hospital René Dubos - Pontoise
Locations (5):
- France (5):
  - Geriatric Department - CHRU Brest, Brest
  - Geriatric Department - CH Cholet, Cholet
  - Geriatric Department - Hospital Louis Mourier - Colombes, Colombes
  - Geriatric Department - Intercommunal hospital center - Créteil, Créteil
  - Geriatric Department - Hospital René Dubos - Pontoise, Pontoise